CLINICAL TRIAL: NCT02108470
Title: A Randomized Cross-over Clinical Trial to Evaluate the Use of Oral Health-Related Quality of Life in Dental Practice
Acronym: OHRQoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: The University of Hong Kong (Other); Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Roslan Saub, Associate Professor, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: ER020-2012A
Record Dates: First submitted 2014-03-31; First posted 2014-04-09 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Oral Health; Quality of Life
Keywords: Oral Health Related Quality of Life (OHRQoL); Oral Health Impact Profile (OHIP); Dentist-Patient Relations; patients' participation.; patients' satisfaction with the consultation.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dental consultation without OHQoL assessment (No Intervention): Dentist performs consultation in the traditional method
- Dental consultation using OHIP (Experimental): Dental consultation using OHIP incorporating OHRQoL issues.
  Interventions: Other: Dental consultation using OHIP

INTERVENTIONS:
Other: Dental consultation using OHIP — The S-OHIP[M] measure assesses the impact of one's oral health condition on QoL, contributing to 7 domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Responses of each item are made on a Likert scale and coded as: 1 = never, 2 =hardly ever, 3= occasionally, 4= fairly often, and 5= very often.
  Other Names: Oral Health Impact Profile (OHIP-14)
  Arms: Dental consultation using OHIP

SUMMARY:
The aim of this study is to determine whether by incorporating an Oral Health-Related Quality of Life (OHRQoL) measure in dental practice will improve patient-dentist communication and enhance patient's satisfaction. The objectives of this study are: (i) To determine the measurement equivalence of Computer Touch Screen Assessment (CTSA) and Paper Based Assessment (PBA) of the Oral Health Impact Profile (OHIP-14). (ii) To evaluate and compare how useful a standardized OHRQoL assessment improves patient-dentist communication with regards to number of relevant OHRQoL issues addressed and percentage of most frequently items discussed between the intervention and control groups, assess the patient's active participation between the intervention and control groups and enhances patient's satisfaction between the intervention and control groups.

DETAILED DESCRIPTION:
The Oral Health Division of the Ministry of Health in Malaysia recognizes that customer centered/ patient-centered care (PCC) is of key importance in providing quality oral health care to the population. This paradigm shift in health care to 'patients' rather than 'providers' in determining health needs and service outcomes requires a more holistic approach relying on active patient involvement. This in turn has led to the development and use of patient-centred health status measures - termed 'health-related quality of life' [HRQoL] within medicine. These HRQoL have proved effective in understanding patients' health needs, ability to cope with illnesses, compliance with treatment and ultimately the overall success of care, thus ensuring PCC. In dentistry, considerable advances have been made in developing valid and reliable HRQoL for oral health [OHRQoL] . The most widely used and sophisticated measures being the Oral health Impact Profile which has been adapted for use and validated in Malaysia. The challenge now is to determine how effective such a measure is in attaining the goal of PCC for dentistry in Malaysia.

Method. This study id divided into two phase; phase 1 & phase 2.

Phase 1; Testing the measurement equivalence of 'Touch-screen' versus 'Paper-based' assessments of OHRQoL:

* Study design: This study is a randomized crossover study design.
* Study Area: Selangor
* Sample and Sampling method:

  * The participants from the residential colleges at a university campus will be randomly assigned through block randomization in groups of four (ABBA) into two arms of the trial:

    (i) Arm A where participants self-completed the CTSA followed by the PBA or (ii) Arm B where participants self-completed PBA followed by CTSA. Intervention (test): The participants answered the Oral Health Impact Profile (OHIP-14) questionnaire using the CTSA.

Standard Protocol (Control): The participants answered the OHIP-14 using the PBA.

Procedure:

1. The participants were randomized to either (i) Arm A: completed CTSA then PBA of OHIP-14, or (ii) Arm B: PBA and then CTSA of OHIP-14 within the same day. User preference and time taken to complete the assessments were recorded. The first assessment was conducted in the morning (AM) session and the second assessment was conducted in the afternoon (PM) session. The period of 'washout' was a 'lunch period' between morning and afternoon sessions.
2. Participants who able to read and speak Malay are eligible to participate in this study.

Data Collection:

1. All eligible participants, who fulfilled the inclusion criteria, will be invited to participate in this study. Assignment to trial arm was concealed in envelopes that were opened when informed consent was obtained from participants.
2. PBA involved 'pen and paper' for participants to self-complete questions. Data from PBA were entered manually into the computer package of SPSS for the analyses.
3. For the CTSA a Samsung tablet with Android operating system was used. The respondents entered their responses by touching the relevant buttons on the screen. The navigation buttons at the bottom of the screen allowed the screen to be moved backwards and forwards through the questions. The responses were compiled automatically into an excel file that could be accessed in Statistical Program for the Social Sciences software (SPSS).
4. The formats of the questions were similar in both CTSA and PBA. The time taken for participants to complete PBA and CTSA was recorded by stopwatch. On completion of the trial participants were asked to rate their preference for PBA or CTSA (touch screen, paper, or no preference).

Phase 2; To evaluate and compare how useful a standardized OHRQoL assessment improves patient-dentist communication :

* Study design: This study is a randomized crossover study design.
* Study Area: Selangor
* Sample and Sampling method:

  * The Community Health Care Centers (CHCC) will be randomized into two groups:

group A and B.

* Group A will start with intervention (test) and follow by the standard protocol (Control) and vice versa for group B.

Intervention (test): Dental consultation will be carried out by incorporating an OHQoL assessment. The OHQoL will be measured globally using Oral Health Impact Profile (S-OHIP[M]).

Standard Protocol (Control): Dental consultation will be carried out in a conventional way (without OHQoL assessment).

Procedure:

1. The participating dentist(s) randomized to group "A" will conduct 35 consultations incorporating the OHQoL assessments (i.e. the intervention) on a selected patients and then following a washout period of 1-month will conduct 35 consultations without OHQoL assessments (control). At those CHCC randomized to group 'B' participating dentist(s) will conduct 35 consultations without incorporating OHQoL assessments (control) and then following a washout period of 1-month will conduct 35 consultations with OHQoL assessments.
2. Patients aged 18 and older with presenting complaint of oral pain are eligible to participate in this study.

Data Collection:

1. All eligible patients, who fulfilled the inclusion criteria, will be invited to participate in this study. Screening for eligibility will be done at the registration site. All patients in the intervention group will be asked to complete the S-OHIP[M] on the touch screen Samsung tablet with Android operating system prior to the consultation. The program will systematically summarize the results of the questionnaire.
2. Dentists in the intervention group will perform the consultation with an addition of using the OHRQoL information as presented on the iPad screen in the consultation.

Dentists in the control group, on the other hand, will perform the conventional consultation. The consultation will be audiotape. At the end of the treatment, patients will be given the satisfaction questionnaire to be completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older with presenting complaint of oral pain are eligible to participate in this study.

Exclusion Criteria:

* Patients who are illiterate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The number or percentage of relevant OHRQoL issues addressed | 1 day ( after dental consultation)
  For each consultation, score will be given based on the number of problems discussed. The composite score can range from 0-14; where 0 no issue discussed and 14 all issues discussed.
The patient's participation between the intervention and control groups | 1 day ( after dental consultation)
  Patient's participation will be measured by determining the length of time patient speaks to the dentist. Estimated duration will be made based on the audiotape.
9-item Consultation Satisfaction Questionnaire (CSQ) will be used in this study. | 1 day ( after dental consultation)
  The CSQ-9 looks at 4 different areas of satisfaction; general satisfaction (2 questions), professional care (4 questions), depth of relationship (2 questions) and perceived time (1 questions).

CONTACTS AND LOCATIONS:
Overall Officials: Roslan Saub, PhD, Principal Investigator — University of Malaya; Colman McGrath, PhD, Principal Investigator — The University of Hong Kong; Zainab Shamdol, Master, Principal Investigator — Ministry of Health, Malaysia
Locations (1):
- Goverment Dental Clinics, Shah Alam, Selangor, Malaysia